CLINICAL TRIAL: NCT06607835
Title: A Preliminary Study Looking at the Use of Cannabis Suppositories and Mindful Compassion Online Groups for Sexual Functioning Among Women Post Gynaecological Cancer Treatment
Brief Title: Cannabis Suppositories and Mindful Compassion Online Groups for Sexual Functioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Metropolitan University (Other)
Responsible Party: Principal Investigator, Samantha Banbury, Principal Investigator, London Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: London Met Uni
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Sexual Pain Disorders
Keywords: mindful-compassion; well-being; sexual self-efficacy; sexual functioning; cannabis suppositories

STUDY DESIGN:
Intervention Model Description: The study phase is not applicable as whilst cannabis suppositories are part of this research study, participants are not randomised into cannabis groups. Participants would already be using cannabis suppositories for at least one month and are used as part of the individuals sexual intimacy.
  Randomisation was based on whether participants were using cannabis suppositories and consisted of one of four groups, including a cannabis suppository-only group, mindful- compassion only group, a combined mindful-compassion and cannabis suppository group and a care-as-usual group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online mindful-compassion weekly for four weeks (Experimental): Mindful compassion exercises
  Interventions: Behavioral: Mindful- compassion
- Cannabis suppositories and online mindful-compassion for vaginal pain (Experimental): Cannabis suppositories and online mindful-compassion for vaginal pain
  Interventions: Behavioral: Mindful-compassion and cannabis suppositories

INTERVENTIONS:
Behavioral: Mindful- compassion — Online mindful-compassion weekly for four weeks
  Arms: Online mindful-compassion weekly for four weeks
Behavioral: Mindful-compassion and cannabis suppositories — Cannabis suppositories and online mindful-compassion for vaginal pain
  Arms: Cannabis suppositories and online mindful-compassion for vaginal pain

SUMMARY:
Research aim: To determine how an online mindful-compassion intervention adjunct with cannabis suppositories might reduce vaginal pain during sexual intimacy among women post-gynaecological cancer treatment. Outcomes are also hoped to increase sexual functioning, well-being, sexual self-efficacy and quality of life.

Research intention: If the combined mindful compassion and cannabis suppository intervention reduces vaginal pain and supports sexual and general well-being, then this research would be repeated on a larger scale targeting psychosexual services.

A brief overview of the intervention:

Mindfulness has been anecdotally discussed in reducing symptoms of vaginal pain and increasing overall well-being. A novel approach to pain management includes medical cannabis, which can be cannabidiol, tetrahydrocannabinol or both. Vaginal suppositories do not create a euphoric high in the same way as oral use, including inhalation.

Quantitatively, randomisation will be based on whether participants use cannabis suppositories or not. This study does not randomise to cannabis groups owing to the legalities in the United Kingdom. Participants included eighty-three consenting participants. Of these, forty-one were using cannabis suppositories. The intervention was delivered for one month, and the follow-up was at twelve weeks. Qualitatively, participants were asked approximately eight open-ended feedback questions throughout the study.

DETAILED DESCRIPTION:
Research looking at mindfulness-based interventions or the use of medical cannabis to support sexual pain is limited, and often, sexual pain goes unreported, which might lead to compromised psychological well-being. Additionally, sexual problems associated with pain and related emotional suffering are frequently overlooked in patients with sexual pain, particularly among those who are post cancer treatments. This research aims to establish the effectiveness of an online mindful compassion intervention adjunct with cannabis suppositories to help minimise sexual pain and increase well-being. This research decided to deliver mindful compassion online because it would economically target a more comprehensive and diverse group. This preliminary study examined how a mindful compassion intervention combined with cannabis suppositories might help minimise sexual pain whilst improving sexual function, well-being, sexual self-efficacy and quality of life.

The main exercises included mindfulness, breathing, relaxation techniques, Mindfulness of the senses and body, and understanding the self. These exercises incorporated the three-model system of emotions, how to attend to the cognitive and physical patterns associated with painful sex, and towards acceptance and self-compassion with fewer symptoms. The mindful-compassion intervention included psychosexual education and vaginal pain, the three-model system of emotions and sexual pain, practising mindful compassion and graded practice and self-care, efficacy, and the relationship with anatomy.

Homework exercises, including education, training, modelling, and enablement, were encouraged. Feedback and support, along with discussing the educational components, training, modelling, and enablement, were addressed throughout this study.

The development of mindful compassion intervention has been based on a taxonomy of behavioural change techniques. This has been used because the taxonomy of behavioural change techniques has been rigorously tested to evidence the effectiveness in supporting interventions associated with change behaviour. The 93 behaviour change techniques are the active ingredients of behaviour change, and each intervention is likely to consist of more than one behaviour change technique and serve as having more than one function. The intervention in this study included twelve domains, of which twenty-three out of the 93 behaviour change techniques listed in the behavioural change technique taxonomy were identified. The selection of these domains used a triangulation process to ensure consistency in mapping the behaviour change techniques to the intervention.

Randomisation was based on whether participants were already using cannabis suppositories or not. Those who did use cannabis suppositories as part of their sex life would have been doing so for at least a month. There was a total of four groups, including a cannabis suppository-only group, a mindful-compassion-only group, a combined mindful compassion and cannabis suppository group and a care-as-usual group.

ELIGIBILITY:
Inclusion Criteria:

* Participants were allocated to cannabis only, and cannabis adjunct groups would already be using cannabis suppositories.
* Must have engaged in vaginal sex within the last month
* Must be at least 6 months post cancer treatment
* Must be based in the United Kingdom
* Must have experienced sexual pain
* An absence of co-occurring difficulties
* Must be aged 18 years or older
* Must be able to read and write English.
* Patient health screening score must range between 0-9 mild
* Generalised anxiety disorder screening score must range between 0-9, mild

Exclusion Criteria:

* Have not attempted vaginal intercourse in the last month
* Have co-occurring difficulties
* Are still receiving cancer treatment or within 6 months of cancer treatment such as chemotherapy, surgery or radiation
* Aged below 18 years old
* Reading and writing English difficulties
* Not experiencing pain during vaginal sexual intercourse.
* Patient health screening score ranged between moderate to severe - 10-27
* Generalised anxiety screening score ranged between 10- 21.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-07-02 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
The Short Warwick -Edinburgh Mental Well-being Scale | 0, 4 and 12 weeks
  This is a 7 item questionnaire with 5 response categories looking at functioning and feeling aspects of well-being. The response categories include 1=none of the time to 5=all of the time. Cronbach alpha for the questionnaire is 0.89-0.91. There is no reverse scoring. Scores range from 7 to 35 where the latter is the highest level of wellbeing. The Cronbach alpha in this study was 0.85.
State Self-compassion Short Form | 0, 4 and 12 weeks
  This is a 12 item measure with 5 response categories, 1 = almost never to 5 = almost always, with higher scores indicating higher levels of self-compassion. The questionnaire measures self-kindness versus. Self-judgement, common humanity versus isolation and mindfulness versus over-identification with painful thoughts and emotions. Reliability Cronbach alpha range between 0.68 and 0.78. The Cronbach alpha in this study was 0.73.
The Female Sexual Function Index | 0, 4 and 12 weeks
  This is a 19 item measure of sexual pain, sexual desire, orgasm, lubrication, and sexual satisfaction with five response categories. The score range is 2.0 to 36.0 with 26.0 being the cut of for sexual dysfunction. Example questions include, Over the past 4 weeks, how often did you experience discomfort or pain during vaginal penetration? and Over the past 4 weeks, how would you rate your level of discomfort or pain during or following vaginal penetration? Cronbach alpha for this questionnaire is .820 and higher. For the present study, the Cronbach alpha was .750.
Sexual Self-Efficacy Scale for Female Sexual Functioning | 0, 4 and 12 weeks
  This is a 37 item measure which embraces aspects of female sexuality such as arousal, desire, orgasm, pain and satisfaction. This is a 10 response category. The score ranges of 0 to10, 11 to 20, and 21 to 30 and represent low, moderate, and high self-efficacy levels. Example questions include anticipating, thinking about, having intercourse without fear or anxiety and Engaging in intercourse without pain or discomfort. The Cronbach alpha is .930 for this questionnaire. For the present study, the Cronbach alpha was .852
Brief Quality of Life Scale | 0, 4 and 12 weeks
  An 8 item questionnaire with five response categories looking at satisfaction with self, friends, family and creativity. This scale is scored by transforming the individual item scores from a 1 to 5 scale to a 0 to 100 scale. Example responses include how I view my life as necessary for my quality of life, and I am satisfied with my friends and friendship: The Cronbach alpha is .760 for this questionnaire. For the present study, the Cronbach alpha was .789.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Banbury, PhD, Principal Investigator — London Metropolitan University
Locations (1):
- School of Social Sciences and Professions, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brotto LA, Yule M, Breckon E. Psychological interventions for the sexual sequelae of cancer: a review of the literature. J Cancer Surviv. 2010 Dec;4(4):346-60. doi: 10.1007/s11764-010-0132-z. Epub 2010 Jul 3. PMID 20602188
- [Result] Brotto LA, Erskine Y, Carey M, Ehlen T, Finlayson S, Heywood M, Kwon J, McAlpine J, Stuart G, Thomson S, Miller D. A brief mindfulness-based cognitive behavioral intervention improves sexual functioning versus wait-list control in women treated for gynecologic cancer. Gynecol Oncol. 2012 May;125(2):320-5. doi: 10.1016/j.ygyno.2012.01.035. Epub 2012 Jan 28. PMID 22293042
- [Result] Brotto LA, Stephenson KR, Zippan N. Feasibility of an Online Mindfulness-Based Intervention for Women with Sexual Interest/Arousal Disorder. Mindfulness (N Y). 2022;13(3):647-659. doi: 10.1007/s12671-021-01820-4. Epub 2022 Jan 4. PMID 35035598
- [Result] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Result] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Result] Libman E, Rothenberg I, Fichten CS, Amsel R. The SSES-E: a measure of sexual self-efficacy in erectile functioning. J Sex Marital Ther. 1985 Winter;11(4):233-47. doi: 10.1080/00926238508405450. PMID 4078907